CLINICAL TRIAL: NCT05615571
Title: Testing of NBIA Genes: Analysis of Genetic Heterogeneity and Validation of Mitochondrial Markers for Assessing Causality of Sequence Variants.
Acronym: NBIA MITO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/38
Record Dates: First submitted 2021-07-01; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-09

CONDITIONS: Neurodegeneration With Brain Iron Accumulation (NBIA)
MeSH Terms: conditions — Pantothenate Kinase-Associated Neurodegeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — cutaneous biopsy and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with NBIA who remain without molecular diagnosis: A group of 40 patients with NBIA, who remain without molecular diagnosis
  Interventions: Genetic: Sequencing tests
- Patients with NBIA with identified mutations in genes: A group of patients with 2 frequent forms of NBIA, carrying mutations in genes (already studied in the CHU molecular diagnostic laboratory)
  Interventions: Genetic: Establishment of mitochondrial markers

INTERVENTIONS:
Genetic: Establishment of mitochondrial markers — Establishment of mitochondrial markers from fibroblasts in culture, obtained from a skin biopsy. Establishment of yeast models to show biochemical mitochondrial alterations: introduction of missense variants in the pantothenate kinase yeast gene Cab1 whose deletion is lethal, followed by growth of mutant strains on fermentation and respiratory media.
  Groups: Patients with NBIA with identified mutations in genes
Genetic: Sequencing tests — sequencing tests of a panel of 22 genes (9 already known and 13 new genes) using a dedicated custom capture and a medium throughput sequencing protocol.
  Groups: Patients with NBIA who remain without molecular diagnosis

SUMMARY:
Neurodegeneration with brain iron accumulation (NBIA) represent a group of rare neurodevelopmental diseases, genetically as well as phenotypically heterogeneous.

The diagnosis is based on brain MRI. It is also based on genetic testing. However overlaps exist between the different clinical presentations and the molecular diagnosis may be misinterpreted.

Two main purposes must be addressed to get a better molecular diagnosis: on one hand reaching enough exhaustivity which may be performed with a larger gene panel and next generation sequencing; on the other hand, it is now necessary to validate or infirm the deleterious consequences of variants with the help of functional studies.

DETAILED DESCRIPTION:
Neurodegeneration with brain iron accumulation (NBIA) represent a group of rare neurodevelopmental diseases, genetically as well as phenotypically heterogeneous.

The diagnosis is based on brain MRI. It shows abnormal deposit of iron in the basal ganglia, especially in the globus pallidus and the substance nigra. It is also based on genetic testing. Ten individualized forms are now described. However overlaps exist between the different clinical presentations and the molecular diagnosis may be misinterpreted because of variants, named as variants of unknown signification, whom the pathogenic role is not proven. Approximately half of the clinically relevant cases with iron deposits on brain MRI remain without any molecular deleterious alteration.

Two main purposes must be addressed to get a better molecular diagnosis: on one hand reaching enough exhaustivity which may be performed with a larger gene panel and next generation sequencing; this panel will include new genes and could be enlarged as more genes are identified. On the other hand, it is now necessary to validate or infirm the deleterious consequences of variants with the help of functional studies.

Four major pathways are involved in the pathophysiology of NBIA: iron and lipids metabolisms, mitochondrial metabolism and autophagy.

Considering that biochemical mechanisms inside the mitochodrion are involved in these four pathways, the investigators performed a first test starting from patient's fibroblasts and analyzed the literature in order to define the parameters that could be pertinent as biological markers of NBIA.

Two different groups will be studied :

* A group of NBIA patients without found mutation after sequencing of the gene panel currently used at the university hospital of Bordeaux. Genetic testing will be performed with the help of an alternative method of target enrichment applied to 16 NBIA genes.
* A group of patients with 2 frequent forms of NBIA with identified variants will be analysed to assess the best mitochondrial markers from fibroblasts.

The investigators plan to transfer these new genetic and biochemical strategies to the diagnostic procedures with the support of the french rare disease network in charge of neurodegenerations and the "CARAMMEL" network involved in the diagnosis of mitochondrial diseases.

ELIGIBILITY:
Inclusion Criteria:

* NBIA Patients diagnosed with a pathogenic variation or any variation that could impact gene function (class 4 or 5 according to ACMG criteria) in the following genes: C19ORF12, PANK2, PLA2G6, DCAF17, FA2H, WDR45, FTL, CP and ATP13A2 and whose fibroblasts have been collected at Bordeaux University Hospital for functional analysis during the diagnosis procedure
* NBIA patients without conclusive testing in none of these nine genes and whose DNA has been collected during the diagnosis procedure at Bordeaux University Hospital

Exclusion Criteria:

* Patients without imaging (MRI or scan) signs of NBIA
* Patients without french healthcare insurance

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with NBIA
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Sequencing tests of a panel of 22 genes using a dedicated custom capture and a medium throughput sequencing protocol. | through study completion, an average of 2 years
  Records of coverage (% of designed regions)
Sequencing tests of a panel of 22 genes using a dedicated custom capture and a medium throughput sequencing protocol. | through study completion, an average of 4 years
  Records of depth of sequencing (reads number)

SECONDARY OUTCOMES:
Identification of the dominant form using biochemical analysis in patient's fibroblasts | through study completion, an average of 2 years
  Counting of mitochondria with Voltage-dependent anion channel (VDAC) labeling
Identification of the dominant form using biochemical analysis in patient's fibroblasts | through study completion, an average of 2 years
  Measurements of iron and ferritin cellular levels after iron deprivation and iron loading

CONTACTS AND LOCATIONS:
Overall Officials: Patricia FERGELOT MAURIN, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Talence, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angelini C, Durand CM, Fergelot P, Deforges J, Vital A, Menegon P, Sarrazin E, Bellance R, Mathis S, Gonzalez V, Renaud M, Frismand S, Schmitt E, Rouanet M, Burglen L, Chabrol B, Desnous B, Arveiler B, Stevanin G, Coupry I, Goizet C. Autosomal Dominant MPAN: Mosaicism Expands the Clinical Spectrum to Atypical Late-Onset Phenotypes. Mov Disord. 2023 Nov;38(11):2103-2115. doi: 10.1002/mds.29576. Epub 2023 Aug 21. PMID 37605305